CLINICAL TRIAL: NCT01209585
Title: Study to Evaluate Biomarkers in Blood and Synovial Fluid in Subjects With Rheumatoid Arthritis
Brief Title: A Study to Evaluate BioMarkers in Blood Samples in Subjects With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: CD-IA-INDP-1056
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Rheumatoid Arthritis: Subject must have RA with inflamed joint
  Interventions: Other: Blood samples; Other: Synovial fluid aspiration; Other: Synovial tissue sample
- Osteoarthritis: Subjects must have OA of the knee
  Interventions: Other: Blood samples; Other: Synovial fluid aspiration; Other: Synovial tissue sample
- Pseudo gout: Subjects must have peusdo-gout of knee

INTERVENTIONS:
Other: Blood samples — Subjects will have visits on Days 1, 30 and 120.
  Groups: Osteoarthritis; Rheumatoid Arthritis
Other: Synovial fluid aspiration — Subjects will have visits on Days 1, 30, and 120.
  Groups: Osteoarthritis; Rheumatoid Arthritis
Other: Synovial tissue sample — Subjects will have visits on Days 1, 30, and 120.
  Groups: Osteoarthritis; Rheumatoid Arthritis

SUMMARY:
The purpose of this study is to study the evaluation of blood samples and blood types to identify functional protein in the joints.

DETAILED DESCRIPTION:
Assessment of type I IFN signature in the peripheral blood and activation of type I IFN signaling pathway in synovial fluid (indicating expression of the functional IFN protein in the joints).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 75 years at time of screening.
* Written informed consent and any locally required authorization (eg, HIPAA in the USA), obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
* A diagnosis of: a) Adult onset RA as defined by the 1987 ACR classification criteria (see Appendix 1), with at least 4 tender and 4 swollen joints at screening (Day 1). Tender/swollen joints must be a part of the 28-joint count included in the Disease Assessment Score 28 (DAS28) assessment; b) Osteoarthritis (OA) of the knee or acute pseudogout attack of the knee.
* Age ≥ 16 years at the time of onset of RA or onset of OA, pseudogout.
* Subjects should either not receive oral corticosteroids, or if receiving oral corticosteroids, need to be on a stable dose of oral prednisone (or equivalent) ≤ 10 mg/day for at least 4 weeks prior to screening (Day 1).
* Ability and willingness to complete the study until Day 120 as required by the protocol.

Exclusion Criteria:

* History or current inflammatory joint disease other than RA, OA, or pseudogout (eg, gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other autoimmune disorder (systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, or overlap syndrome).
* Any neurological (congenital or acquired), psychiatric, vascular, or systemic disorder could also affect the evaluation of disease assessments; in particular, joint pain and swelling.
* Treatment with IFN-α or IFN-β.
* Intra-articular, IM, or IV corticosteroid injections within 28 days before screening (Day 1).
* Known history of or positive test result for human immunodeficiency virus (HIV).
* Serious infection (eg, pneumonia, septicemia) within the 2 months prior to Day 1 visit.
* Active bacterial or viral infection (which includes ongoing and/or chronic infections such as hepatitis, tuberculosis, etc).
* Concomitant use of systemic antiviral, antibiotic, or antifungals for the treatment of active infection within 28 days of Day 1.
* History of malignancy or evidence of active or suspected malignancy (with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix > 1 year before randomization into the study).
* Vaccinations within 4 weeks of Day 1 visit.
* Concurrent enrollment in another clinical study.
* Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals.
* Other unspecified reasons that, in the opinion of the Investigator or medical monitor, make the subject unsuitable for participation or confound the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or Female Adults aged 18-75 years old
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Data Collection and Analyses | Study Day 120
  Data analyses on model devlopment to maximize measures of predictive diagnostic accuracy, etc.

SECONDARY OUTCOMES:
RNA Assessment | Day 120
  Level of signature protein, messenger RNA or micro RNA in peripheral blood and diseased tissue will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Warren Greth, MD, Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Research Site, Frederick, Maryland
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Jackson, Tennessee